CLINICAL TRIAL: NCT00124917
Title: A Phase I Study of Image Guided Dose Escalation With Intensity Modulated Radiation Therapy (IMRT) to Histologically Confirmed Regions of Prostate Cancer
Brief Title: Phase I Study of Intensity Modulated Radiation Therapy for Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to unanticipated toxicity/risks to subjects.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050191; 05-C-0191; NCT00227799 (obsolete NCT alias)
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; Fiducial Marker; IMRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy (Experimental): Radiation to tumor area as per protocol
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Areas of pathologically confirmed malignancy will undergo dose escalation as described below. Areas of image abnormality that could not be biopsied or were without definite pathologic evidence of malignancy will be given intermediate doses. The remainder of the prostate gland will receive standard dose (as per the Radiation Therapy Oncology Group (RTOG) 9406 study) 7560 centigray (cGy) in 180 cGy daily fractions.[1]

SUMMARY:
BACKGROUND:

-This study represents a progression from findings in four previous National Cancer Institute (NCI) Radiation Oncology Branch (ROB) protocols (02-C-0167A, 02-C-0207E, 03-C-0190B, 04-C-0171). In these previous works we have begun to develop techniques to obtain magnetic resonance (MR) biological images and co-register tissue in prostate cancer patients.

OBJECTIVES:

-The scientific objective of this protocol is to determine the maximum tolerated dose (MTD) of external beam radiation to regions of interest within the prostate based acute toxicity.

Secondary objectives of this study are to relate patterns in gene and protein expression to response and toxicity and to evaluate the frequency of late term toxicity.

ELIGIBILITY:

-Patients with prostate cancer without evidence of metastasis will be eligible for this study.

DESIGN:

* This phase I trial will use intensity modulated radiation therapy (IMRT) to deliver escalating doses of external beam radiation to regions of histologically confirmed prostate cancer. The study will be conducted using a standard 3-6 dose-escalation with an initial 3 patients in each dose cohort and the potential expansion of the cohort to 6 patients.
* Anatomic magnetic resonance imaging (MRI) and magnetic resonance (MR) biological images, such as magnetic resonance spectroscopy (MRS), will be obtained. Tissue will be acquired from sites of interest, with biopsy locations precisely translated (co-registered) to an MR image of reference. Tissue samples will be processed for complementary deoxyribonucleic acid (cDNA) microarray testing and stored for future analysis in the Radiation Oncology Branch, NCI. A gold seed will be left at the biopsy site as a fiducial marker to direct future radiation therapy. If necessary, additional fiducial markers will be placed for target localization during treatment.
* Once MR guided biopsies are obtained and fiducial markers placed, the patient will undergo a standard computed tomography (CT) simulation for radiation therapy treatment planning. The MR and CT images will be fused. Areas of pathologically confirmed malignancy will undergo dose escalation as described below. Areas of image abnormality that could not be biopsied or were without definite pathologic evidence of malignancy will be given intermediate doses. The remainder of the prostate gland will receive standard dose (7560 centigray (cGy)').
* The trial will accrue 18 to 36 patients with an anticipated accrual period of 2 years.

DETAILED DESCRIPTION:
BACKGROUND:

-This study represents a progression from findings in four previous National Cancer Institute (NCI) Radiation Oncology Branch (RO)B protocols (02-C-0167A, 02-C-0207E, 03-C-0190B, 04-C-0171). In these previous works we have begun to develop techniques to obtain magnetic resonance (MR) biological images and co-register tissue in prostate cancer patients.

OBJECTIVES:

* The scientific objective of this protocol is to determine the maximum tolerated dose (MTD) of external beam radiation to regions of interest within the prostate based acute toxicity.
* Secondary objectives of this study are to relate patterns in gene and protein expression to response and toxicity and to evaluate the frequency of late term toxicity.

ELIGIBILITY:

-Patients with prostate cancer without evidence of metastasis will be eligible for this study.

DESIGN:

* This phase I trial will use intensity modulated radiation therapy (IMRT) to deliver escalating doses of external beam radiation to regions of histologically confirmed prostate cancer. The study will be conducted using a standard 3-6 dose-escalation with an initial 3 patients in each dose cohort and the potential expansion of the cohort to 6 patients.
* Anatomic magnetic resonance imaging (MRI) and MR biological images, such as magnetic resonance spectroscopy (MRS), will be obtained Tissue will be acquired from sites of interest, with biopsy locations precisely translated (co-registered) to an MR image of reference. Tissue samples will be processed for complementary deoxyribonucleic acid (cDNA) microarray testing and stored for future analysis in the Radiation Oncology Branch, NCI. A gold seed will be left at the biopsy site as a fiducial marker to direct future radiation therapy. If necessary, additional fiducial markers will be placed for target localization during treatment.
* Once MR guided biopsies are obtained and fiducial markers placed, the patient will undergo a standard computed tomography (CT) simulation for radiation therapy treatment planning. The MR and CT images will be fused. Areas of pathologically confirmed malignancy will undergo dose escalation as described below. Areas of image abnormality that could not be biopsied or were without definite pathologic evidence of malignancy will be given intermediate doses. The remainder of the prostate gland will receive standard dose (7560 centigray (cGy)).
* The trial will accrue 18 to 36 patients with an anticipated accrual period of 2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
  2. Pathology report confirming adenocarcinoma of the prostate
  3. Risk of lymph node metastasis less than 10% as defined by the Partin tables
  4. Tumor visible on magnetic resonance imaging (MRI)
  5. No prior surgery, radiation, or chemotherapy for prostate cancer.
  6. Age greater than 18 y/o and less than 90 years old.

EXCLUSION CRITERIA:

1. Cognitively impaired patients who cannot give informed consent.
2. Patients with metastatic disease.
3. Contraindication to biopsy

   * Bleeding disorder
   * Prothrombin time (PT)/Partial Thromboplastin Time (PTT) greater than or equal to 1.5 times the upper limit of normal
   * Platelets less than or equal to 50K
   * Artificial heart valve
4. Contraindication to magnetic resonance imaging (MRI)

   * Patients weighing greater than 136 kgs (weight limit for the scanner tables)
   * Allergy to MR contrast agent
   * Patients with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices.
5. Pre-existing and active prostatitis or proctitis
6. Other medical conditions deemed by the principal investigator (PI) or associates to make the patient ineligible for protocol investigations, procedures, and high-dose external beam radiotherapy.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-07-21 (Actual); Primary Completion 2011-03-06 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aradhana Kaushal, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michalski JM, Winter K, Purdy JA, Perez CA, Ryu JK, Parliament MB, Valicenti RK, Roach M 3rd, Sandler HM, Markoe AM, Cox JD. Toxicity after three-dimensional radiotherapy for prostate cancer with RTOG 9406 dose level IV. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):735-42. doi: 10.1016/S0360-3016(03)01578-5. PMID 14967428
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Pollack A, Hanlon A, Horwitz EM, Feigenberg S, Uzzo RG, Price RA. Radiation therapy dose escalation for prostate cancer: a rationale for IMRT. World J Urol. 2003 Sep;21(4):200-8. doi: 10.1007/s00345-003-0356-x. Epub 2003 Sep 5. PMID 12961097

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 6 participants enrolled in this trial received a dose of 7560 cGy and are grouped together in one Arm/Group. An attempt was made to escalate to the next higher dose but we were unable to treat patients and maintain safety standards.
Groups:
- Radiation Therapy - 7560 cGY: Radiation to tumor area as per protocol
  Radiation: Areas of pathologically confirmed malignancy will undergo dose escalation as described below. Areas of image abnormality that could not be biopsied or were without definite pathologic evidence of malignancy will be given intermediate doses. The remainder of the prostate gland will receive standard dose (as per the Radiation Therapy Oncology Group (RTOG) 9406 study) 7560 centigray (cGy) in 180 cGy daily fractions.[1]
Period: Overall Study
Arm/Group | Radiation Therapy - 7560 cGY
Started | 6
Completed | 3
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: All 6 participants enrolled in this trial received a dose of 7560 cGy and are grouped together in one Arm/Group. An attempt was made to escalate to the next higher dose but we were unable to treat patients and maintain safety standards.
Arm/Group | Radiation Therapy - 7560 cGY
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.17 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of External Beam Radiation
Description: Maximum tolerated dose is defined as the dose level immediately below the dose level at which 2 or more in a cohort of either 3 or 6 patients experienced a dose limiting toxicity attributed to radiation therapy.
Time Frame: 12 weeks after radiation therapy (RT)
Population: This outcome measure was not done. All 6 participants enrolled in this trial received a dose of 7560 cGy and are grouped together in one Arm/Group. An attempt was made to escalate to the next higher dose but we were unable to treat patients and maintain safety standards.
Arm/Group | Radiation Therapy - 7560 cGY
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTC v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 53 months and 20 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy - 7560 cGY
Number analyzed (Participants) | 6
Participants | 3

3. Other Pre Specified Outcome: Radiation Response With Genomic and Proteomic Analyses
Description: Genomic and proteomic analyses will be conducted on a gene by gene basis using a 2-sample t-test at the 0.001 level and correlated with radiation response.
Time Frame: completion of therapy
Population: This outcome measure was not done because the study was closed due to unanticipated toxicity and risks to subjects.
Arm/Group | Radiation Therapy - 7560 cGY
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Correlate Toxicity With Genomic and Proteomic Analyses
Description: Genomic and proteomic analyses will be conducted on a gene by gene basis using a 2-sample t-test at the 0.001 level and correlated with toxicity.
Time Frame: Completion of therapy
Population: This outcome measure was not done because the study was closed due to unanticipated toxicity and risks to subjects.
Groups:
- Radiation Therapy - 7560 cGY: Radiation to tumor area as per protocol
  Radiation: Areas of pathologically confirmed malignancy will undergo dose escalation as described below. Areas of image abnormality that could not be biopsied or were without definite pathologic evidence of malignancy will be given intermediate doses. The remainder of the prostate gland will receive standard dose (as per the Radiation Therapy Oncology Group (RTOG) 9406 study) 7560 centigray (cGy) in 180 centigray (cGy) daily fractions.[1]
Arm/Group | Radiation Therapy - 7560 cGY
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Long-term Effects and Toxicity Following Selective Intra-prostatic Dose Escalation
Description: Acute and late toxicity will be assessed by the Radiation Therapy Oncology Group (RTOG) Acute and Late Toxicity Genitourinary (GI)/Gastrointestinal (GU) scales.
Time Frame: completion of therapy
Population: This outcome measure was not done because the study was closed due to unanticipated toxicity and risks to subjects.
Arm/Group | Radiation Therapy - 7560 cGY
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 53 months and 20 days
Description: All 6 participants enrolled in this trial received a dose of 7560 cGy and are grouped together in one Arm/Group. An attempt was made to escalate to the next higher dose but we were unable to treat patients and maintain safety standards.
Arm/Group | Radiation Therapy - 7560 cGY
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy - 7560 cGY (N=6)
Mood alteration:: Depression (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy - 7560 cGY (N=6)
Bladder spasms (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ejaculatory dysfunction (Reproductive system and breast disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Gastrointestinal - Other (Bloody stools) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Hemorrhoids) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Loose stools) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Loose stools, urgency) (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 1 (2)
Incontinence, urinary (Renal and urinary disorders) | 1 (2)
Libido (Reproductive system and breast disorders) | 2 (2)
Mood alteration::Depression (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain - Other (Generalized body) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (Lower back) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain::Penis (Reproductive system and breast disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Renal/Genitourinary - Other, Dysuria (Renal and urinary disorders) | 3 (5)
Renal/Genitourinary - Other, Weak stream (Renal and urinary disorders) | 2 (4)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (5)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (2)
Weight gain (General disorders) | 3 (4)
Weight loss (General disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT00124917/Prot_SAP_000.pdf
  • Informed Consent Form (2009-04-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT00124917/ICF_001.pdf